CLINICAL TRIAL: NCT06143397
Title: Effect of Transcutaneous Posterior Tibial Nerve Stimulation and Parasacral Transcutaneous Electrical Stimulation on Neurogenic Overactive Bladder Symptoms in Female Patients With Multiple Sclerosis.
Brief Title: Effect of TTNS and PNS on Neurogenic Overactive Bladder Symptoms in Female Patients With Multiple Sclerosis.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization (Other)
Collaborators: Marmara University (Other)
Responsible Party: Principal Investigator, Busra Aydin Erkilic, Physiotherapist, Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Neurogenic Bladder
Record Dates: First submitted 2023-11-16; First posted 2023-11-22 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Multiple Sclerosis; Overactive Bladder Syndrome
MeSH Terms: conditions — Multiple Sclerosis | interventions — Behavior Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The statistician will be blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- TTNS (Transcutaneous tibial nerve stimulation) (Experimental)
  Interventions: Device: TTNS (Transcutaneous tibial nerve stimulation); Behavioral: Behavioral treatment
- PNS (Parasacral nerve stimulation) (Experimental)
  Interventions: Device: PNS (Parasacral nerve stimulation); Behavioral: Behavioral treatment
- Sham stimulation (Sham Comparator)
  Interventions: Device: Sham stimulation; Behavioral: Behavioral treatment

INTERVENTIONS:
Device: TTNS (Transcutaneous tibial nerve stimulation) — Electrodes will be placed in two areas simultaneously (posterior tibial nerve and parasacral locations). Only the electrodes going to the tibial region will be activated, the parasacral electrodes will not be active. A Biolito (MTR+Vertriebs GmbH, Berlin) stimulator will be used to perform posterior tibial nerve stimulation. Stimulation will be delivered via two 50 mm x 50 mm adhesive electrode pads under the left medial malleolus and 5 cm proximal to the distal electrode. Appropriate electrode site will be confirmed by the presence of big toe plantar flexion during stimulation (stimulus intensity will be adjusted according to the patient's tolerance for 200 μs duration at 10 Hz frequency). Stimulation will be applied 2 days a week, each application for 30 minutes, for 6 weeks.
  Arms: TTNS (Transcutaneous tibial nerve stimulation)
Device: PNS (Parasacral nerve stimulation) — Electrodes will be placed in two areas simultaneously (posterior tibial nerve and parasacral locations). Only the electrodes going to the parasacral region will be activated, the tibial electrodes will not be active. For parasacral region stimulation, electrodes will be positioned symmetrically in the parasacral region under the posterior superior iliac spines to stimulate the S2 and S3 nerve roots. A duration of 200 μs at a frequency of 10 Hz will be set with the Biolito (MTR+Vertriebs GmbH, Berlin) stimulator. The intensity level will be adjusted according to the tolerance of the patient. Stimulation will be applied 2 days a week, each application for 30 minutes, for 6 weeks.
  Arms: PNS (Parasacral nerve stimulation)
Device: Sham stimulation — Electrodes will be placed in three areas simultaneously. These regions are the tibial and parasacral locations and the scapular region, with a distance of approximately 4 cm between the electrodes. Of these three regions, only the channel to the scapular region will be activated, the remaining two regions will be closed. Regarding the sham group, the parameters used in the scapular region will be applied with a frequency of 100 Hz, a pulse duration of 100 μs, and 30 minutes. This configuration is known as conventional transcutaneous electrical nerve stimulation and is commonly used for non-invasive and non-pharmacological treatment of pain.Stimulation will be applied 2 days a week, each application for 30 minutes, for 6 weeks.
  Arms: Sham stimulation
Behavioral: Behavioral treatment — It includes techniques and skills to prevent incontinence and restrain the urge to urinate. It also includes lifestyle interventions such as losing weight, relieving constipation, quitting smoking, reducing caffeine, managing uric acid, wearing non-restrictive, easily removable clothing, reducing emotional stress, and correcting faulty frequent urination by introducing avoidance and distraction techniques. Additionally, advice on proper voiding position and an exercise protocol will be given. The exercise protocol will include three sets of 8-10 near-maximal contractions in lying, sitting and standing positions. Each contraction will be based on the endurance of the pelvic floor muscles and the participant will aim to hold the muscles for 10 seconds. They will be told to do it twice a day, morning and evening. Participants will perform the behavioral training protocol at home.

SUMMARY:
This study aims to evaluate the use of transcutaneous tibial nerve stimulation (TTNS) and parasacral nerve stimulation (PSS) methods in the treatment of overactive bladder (OAB) symptoms in patients with Multiple Sclerosis (MS), including urination frequency, urgency, urinary incontinence, post-void residue, maximum micturition rate. To investigate the effect on parameters such as voiding volume and quality of life and to compare the final results between groups.

DETAILED DESCRIPTION:
Participants will be divided into 3 groups: TTNS, PNS, and placebo groups, and all participants will be given behavioral treatment. Tibial nerve stimulation will be given to the TTNS group, sacral nerve stimulation will be given to the PNS group, and sham current will be given to the placebo group. Stimulation treatments will be applied 2 days a week for 30 minutes each for 6 weeks. Participants will be evaluated before and after treatment. The parameters of urination frequency, urgency, and urinary incontinence will be evaluated with a 3-day voiding diary (BD), maximum flow rate (Qmax), time to reach maximum flow (TQmax), average flow rate, flow time (Tw), voiding time and voiding volume (VV) values will be evaluated by uroflowmetry, post-voiding residual (PVR) volume will be evaluated by ultrasound, and quality of life will be evaluated by King's Quality of Life Questionnaire (KHQ); Expanded Disability Status Scale (EDSS), Overactive bladder form (OAB-v8), Incontinence Severity Index (ISI), Neurogenic Bladder Symptom Score (NBSS) will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Having symptoms related to overactive bladder (OAB-v8 score ⩾8),
* Over 18 years of age
* No relapse for at least 1 month
* All types of MS, including those with relapses
* Female MS patients with an Expanded Disability Status Scale (EDSS) score below 7.0
* Agreeing to participate in the research

Exclusion Criteria:

* Patients with urinary tract infections
* Patients diagnosed with diabetes mellitus
* Patients using diuretic drugs or patients with a clean intermittent catheter
* Patients with a history of different urological diseases
* Patients with heart or brain pacemaker users, those with epilepsy, and patients with language and cognitive limitations
* Patients who are pregnant or in the postpartum period
* Lack of activity performance for 2 weeks (regardless of which group)

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2023-11-20 (Actual); Primary Completion 2025-10-20 (Actual); Study Completion 2025-10-30 (Actual)

PRIMARY OUTCOMES:
Uroflowmetry | Baseline
  It provides a valuable non-invasive assessment of voiding functions. It is the measurement of urine flow rate in ml/sec with the help of a flow meter. Since it is non-invasive among urodynamic tests, it can be used for screening purposes. Pattern and rate of flow depend on detrusor function and bladder outlet resistance.
Uroflowmetry | After the 6-week intervention
  It provides a valuable non-invasive assessment of voiding functions. It is the measurement of urine flow rate in ml/sec with the help of a flow meter. Since it is non-invasive among urodynamic tests, it can be used for screening purposes. Pattern and rate of flow depend on detrusor function and bladder outlet resistance.
Post voiding residue (PVR) | Baseline
  PVR will be measured using a 5-13-MHz convex ultrasound probe.
Post voiding residue (PVR) | After the 6-week intervention
  PVR will be measured using a 5-13-MHz convex ultrasound probe.

SECONDARY OUTCOMES:
Overactive bladder form (OAB-v8) | Baseline
  OAB-v8 is an eight-item screening test for overactive bladder (OAB) symptoms and has been validated in Turkish. The total score is between 0 and 40. Higher scores indicate OAB symptom burden and severity.
Three-day bladder diary (BD) | Baseline
  BD contains the most critical parameters for measuring the frequency and severity of LUTS according to International Continence Society (ICS) recommendations and definitions. The 3-day bladder diary measures the frequency of urination, nocturia, urgency, and urge incontinence for 3 consecutive days. The average frequency of each symptom over three days will be considered the final result.
King's Quality of Life Questionnaire (KHQ) | Baseline
  One of the commonly used quality of life measures for urinary dysfunction is the King's Quality of Life Questionnaire. It is one of the most valid and widely used questionnaires that targets the quality of life in patients with urinary incontinence and precisely measures the impact of urinary incontinence symptoms on the quality of life.
Incontinence Severity Index (ISI) | Baseline
  Developed for use in epidemiological and clinical studies to identify women suffering from urinary incontinence, ISI, used in many different urinary incontinence studies, consists of two questions and the total score obtained by multiplying the frequency of urinary incontinence and the amount of urinary incontinence varies between 1 and 12.
Neurogenic Bladder Symptom Score (NBSS) | Baseline
  The Neurogenic Bladder Symptom Score (NBSS) is a discriminatory tool developed for use in patients with spinal cord injuries, multiple sclerosis, and spina bifida. There are a total of 22 questions covering incontinence, storage and voiding symptoms, as well as urinary complications associated with neurogenic bladder dysfunction.
Overactive bladder form (OAB-v8) | After the 6-week intervention
  OAB-v8 is an eight-item screening test for overactive bladder (OAB) symptoms and has been validated in Turkish. The total score is between 0 and 40. Higher scores indicate OAB symptom burden and severity.
Three-day bladder diary (BD) | After the 6-week intervention
  BD contains the most critical parameters for measuring the frequency and severity of LUTS according to International Continence Society (ICS) recommendations and definitions. The 3-day bladder diary measures the frequency of urination, nocturia, urgency, and urge incontinence for 3 consecutive days. The average frequency of each symptom over three days will be considered the final result.
King's Quality of Life Questionnaire (KHQ) | After the 6-week intervention
  One of the commonly used quality of life measures for urinary dysfunction is the King's Quality of Life Questionnaire. It is one of the most valid and widely used questionnaires that targets the quality of life in patients with urinary incontinence and precisely measures the impact of urinary incontinence symptoms on the quality of life.
Incontinence Severity Index (ISI) | After the 6-week intervention
  Developed for use in epidemiological and clinical studies to identify women suffering from urinary incontinence, ISI, used in many different urinary incontinence studies, consists of two questions and the total score obtained by multiplying the frequency of urinary incontinence and the amount of urinary incontinence varies between 1 and 12.
Neurogenic Bladder Symptom Score (NBSS) | After the 6-week intervention
  The Neurogenic Bladder Symptom Score (NBSS) is a discriminatory tool developed for use in patients with spinal cord injuries, multiple sclerosis, and spina bifida. There are a total of 22 questions covering incontinence, storage and voiding symptoms, as well as urinary complications associated with neurogenic bladder dysfunction.

CONTACTS AND LOCATIONS:
Locations (1):
- Prof.Dr.Cemil Taşcıoğlu Şehir Hastanesi, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Marzouk MH, Darwish MH, El-Tamawy MS, Morsy S, Abbas RL, Ali AS. Posterior tibial nerve stimulation as a neuromodulation therapy in treatment of neurogenic overactive bladder in multiple sclerosis: A prospective randomized controlled study. Mult Scler Relat Disord. 2022 Dec;68:104252. doi: 10.1016/j.msard.2022.104252. Epub 2022 Oct 17. PMID 36274285
- [Background] Jacomo RH, Alves AT, Lucio A, Garcia PA, Lorena DCR, de Sousa JB. Transcutaneous tibial nerve stimulation versus parasacral stimulation in the treatment of overactive bladder in elderly people: a triple-blinded randomized controlled trial. Clinics (Sao Paulo). 2020 Jan 10;75:e1477. doi: 10.6061/clinics/2020/e1477. eCollection 2020. PMID 31939564